CLINICAL TRIAL: NCT06582225
Title: Internet-delivered Cognitive-behaviour Therapy for Obsessive- Compulsive Disorder in Children With Autism: A Randomised Controlled Trial
Brief Title: ICBT for OCD in Children With Autism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Region Skane (Other); Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, David Mataix-Cols, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-01968-01
Record Dates: First submitted 2024-08-28; First posted 2024-09-03 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Obsessive-Compulsive Disorder; Autism Spectrum Disorder
Keywords: Obsessive-Compulsive Disorder; Autism Spectrum Disorder; Exposure and Response Prevention; Cognitive-Behavioural Treatment; Internet; Guided self-help; Stress Management
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Multisite parallel-group randomised controlled superiority trial.
Who Masked: Outcomes Assessor
Masking Description: All study personnel who can be blind to study aims/hypotheses and group allocation, will be blind. Assessors conducting post-treatment and follow-up assessments will be external to the research team and blind to study aims/hypotheses and treatment allocation for the full duration of the trial (up to the 6-month follow-up). The assessors will not receive any information about the study design, objectives or treatment conditions in order to maximise the blinding integrity. At each follow-up assessment, participants will be reminded by their assessor to not reveal details about their treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-delivered exposure and response prevention (I-ERP) (Experimental): A therapist-guided, internet-delivered exposure and response prevention (I-ERP) programme for children and adolescents with OCD and autism.
  Interventions: Behavioral: Internet-delivered exposure and response prevention (I-ERP)
- Internet-delivered stress management (I-SM) (Active Comparator): A therapist-guided, internet-delivered stress management (I-SM) programme for children and adolescents with OCD and autism.
  Interventions: Behavioral: Internet-delivered stress management (I-SM)

INTERVENTIONS:
Behavioral: Internet-delivered exposure and response prevention (I-ERP) — The intervention is internet-delivered and therapist-guided, involving the child and at least one caregiver. It consists of two separate sets of modules, one for the child and one for the caregiver. The intervention consists of 12 modules, delivered over a maximum of 14 weeks.
  The treatment includes psychoeducation about ASD, OCD, emotions, healthy habits, the difference between repetitive behaviours in autism and OCD, how compulsions maintain the obsessions, and the rationale for ERP. The main focus of the treatment is ERP tasks based on the young person's individual goals. The modules also contain homework tasks that are meant to be completed between modules, mainly consisting of ERP. The final module includes a summary of the treatment and a relapse prevention plan.
  The version for parents consists of the same content as the child treatment, but with elaborated psychoeducation, and additional focus on strategies on how to assist their child in the different exposure tasks.
  Arms: Internet-delivered exposure and response prevention (I-ERP)
Behavioral: Internet-delivered stress management (I-SM) — The intervention is internet-delivered and therapist-guided, involving the child and at least one caregiver. It consists of two separate sets of modules, one for the child and one for the caregiver. The intervention consists of 12 modules, delivered over a maximum of 14 weeks.
  The treatment includes psychoeducation about ASD, OCD, healthy habits, and how stress is a contributor to OCD symptoms. The rationale is that targeting and reducing stress will have a beneficial impact on anxiety, obsessions, and compulsions. The main goal of the treatment is to learn how to reduce stress, mainly by using relaxation techniques such as deep breathing, progressive muscle relaxation, and imagery (cognitive) relaxation. The modules also contain homework tasks that are meant to be completed between modules, mainly consisting of relaxation tasks.
  The version for parents contains psychoeducation, as well as strategies on how to assist their child in the different relaxation tasks.
  Arms: Internet-delivered stress management (I-SM)

SUMMARY:
The purpose of this trial is to evaluate the clinical efficacy, the cost-effectiveness and the effect durability of a therapist-guided, internet-delivered cognitive-behavior therapy intervention for obsessive-compulsive disorder (OCD) in children and adolescents with autism. A process evaluation of the treatment will also be conducted.

DETAILED DESCRIPTION:
Primary objective: To determine the clinical efficacy of autism-adapted internet-delivered exposure with response prevention (I-ERP) in reducing OCD symptom severity (as measured by the Children's Yale Brown-Obsessive Compulsive Scale; CY-BOCS) in children and adolescents with OCD and autism spectrum disorder (ASD), compared with an active control intervention of high ecological validity (internet-delivered stress management; I-SM).

Secondary objectives:

1. To establish the 6-month durability of the treatment effects in a naturalistic follow-up.
2. To conduct a health economic evaluation of I-ERP, compared with I-SM, at the primary endpoint (3-month follow-up) from the health organisation payer, health care sector, and societal perspectives.
3. To conduct a process evaluation with a subset of participants allocated to the I-ERP arm, focusing on implementation, mechanisms of impact, and context.

Type of trial: A multisite parallel-group randomised controlled superiority trial, with embedded health economic and process evaluation.

Rationale: OCD and ASD are two frequently co-occuring disorders, associated with significant impairments in daily life. Cognitive-behavioural therapy (CBT) specifically adapted to ASD is a promising treatment for this patient group, but further research is needed to fully establish its efficacy. Furthermore, ASD-adapted CBT for OCD is a highly specialised treatment, not accessible for most patients. Offering treatment in a digital format could dramatically increase treatment availability for these children.

Planned trial sites: The study will be coordinated from the Department of Clinical Neuroscience at Karolinska Institutet (the Sponsor). There will be three collaborating study sites: BUP OCD och relaterade tillstånd (Region Stockholm), BUP Specialmottagning (Västra Götalandsregionen), and BUP Skåne (Region Skåne). Each of the three sites will assess and treat participants from their own region, and occasionally from adjacent regions.

Trial design and methods: All potential participants are initially screened via the telephone or at one of the three participating centres. If screening is positive, an inclusion assessment will follow. Individuals who are eligible and have consented to participate in the trial will be randomised to one of two trial arms. In one arm, participants will receive 12 modules of therapist- and parent-guided I-ERP for OCD adapted for autism. In the active comparator arm, participants will receive 12 modules of therapist- and parent-guided I-SM. Participants in the comparator group will be offered to cross-over to the I-ERP intervention after the primary endpoint.

Participants will complete outcome measures at baseline (week 0), post-treatment (week 12), and 3- and 6-months post-treatment. The primary outcome variable is the clinician-reported Children's Yale Brown-Obsessive Compulsive Scale (CY-BOCS), and the primary endpoint is the 3-month follow-up after treatment.

Secondary outcomes include measures of self-reported OCD symptoms, family accommodation, functional impairment, and depressive symptoms. Health-related quality of life and resource use will be collected for the health economic evaluation. Follow-up assessments will be conducted at the clinic or via videoconferencing, in both cases complemented with online questionnaires.

A subset of participants will participate in a process evaluation of the I-ERP intervention.

Sample: A total of 220 autistic children and adolescents diagnosed with OCD and their primary caregivers.

Statistical methodology and analysis: Data will be analysed using a pre-specified intention-to-treat statistical analysis plan. The primary outcome will be analysed using a linear mixed effects model. Secondary outcomes will be analysed using analogous methods. A health economic evaluation of the intervention from the health organisation payer, health care sector, and societal perspectives will also be conducted, as well as a process evaluation including both quantitative and qualitative measures.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of autism, based on the diagnostic criteria of the 4th or 5th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM) or the 10th edition of the International Classification of Diseases (ICD-10). Informed by the parent/caregiver and subsequently confirmed by review of the medical record or the neurodevelopmental assessment report. A diagnosis of autism will be considered present if it was established with validated instruments, such as the Autism Diagnostic Interview-Revised (ADI-R), the Autism Diagnostic Observation Schedule (ADOS) edition 1 or 2 or the Diagnostic Interview for Social and Communication Disorders (DISCO; autism or ASD cut-offs).
2. A DSM-5 or ICD-10 diagnosis of OCD. Confirmed by the assessor at the inclusion assessment, based on a structured diagnostic interview.
3. A total score of ≥16 on the CY-BOCS. Confirmed by the assessor at the inclusion assessment.
4. Age between 7 and 17 years. Confirmed by the caregiver and subsequently by the medical record system.
5. Ability to read and write Swedish. Confirmed by the caregiver at the telephone screening or/and the inclusion assessment.
6. Regular access to a computer or a smartphone/tablet connected to the internet, and a mobile phone to receive text messages. Confirmed by the caregiver at the telephone screening or/and inclusion assessment.
7. A parent/caregiver able to participate in the treatment alongside their child. Confirmed by the caregiver at the telephone screening or/and the inclusion assessment.

Exclusion Criteria:

1. Global intellectual disability. Informed by the parent/caregiver and subsequently confirmed by review of the medical record or the neurodevelopmental assessment report, and additionally estimated with the two subtests matrix reasoning and similarities from the Wechsler Intelligence Scale for Children - fifth edition (WISC-V) or Wechsler Adult Intelligence Scale - fourth edition (WAIS-IV).
2. Comorbid psychotic disorder, bipolar disorder, severe eating disorder, severe depression, alcohol/substance dependence or hoarding disorder. Confirmed by the caregiver at the telephone screening and subsequently by the assessor at the inclusion assessment based on the structured diagnostic interview and, if required, the medical record.
3. Current suicidal intent or a previous suicide attempt within the last 12 months. Confirmed by the assessor at the inclusion assessment and, if required, the medical record.
4. Main symptom presentation consists of hoarding symptoms. Confirmed by the assessor at the inclusion assessment.
5. Completed CBT for OCD within the last 12 months prior to the inclusion assessment (defined as at least 5 sessions of CBT including ERP). Confirmed by the caregiver at the telephone screening or/and inclusion assessment and, if required, the medical record.
6. Simultaneous psychological treatment for OCD or anxiety. Confirmed by the caregiver at the telephone screening and/or inclusion assessment.
7. Initiation, dosage change or cessation of medication for OCD (primarily selective serotonin reuptake inhibitors, SSRIs) or behavioural symptoms of ASD (atypical antipsychotics) within the 6 weeks prior to the baseline assessment. Confirmed by the caregiver at the telephone screening and the inclusion assessment and, if required, the medical record.
8. Having a close relationship to an already included participant (e.g., sibling, cousin), to avoid being randomised into two different arms, with the risk of information "leaking" between the groups. Confirmed by the caregiver or assessor at the telephone screening and/or at the inclusion assessment.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) | Baseline (week 0), post treatment (week 12), 3-months follow-up, 6-months follow up.
  The CY-BOCS is a semi-structured clinician-administered scale used to assess the severity of OCD symptoms in children and adolescents. The scale consists of a checklist of obsessions and compulsions, 10 items assessing the severity of the OCD symptoms, and a series of ancillary items (e.g., level of insight, avoidance). Range: 0-40, lower scores mean better outcome.

SECONDARY OUTCOMES:
Clinical Global Impression - Severity (CGI-S) | Baseline (week 0), post treatment (week 12), 3-months follow-up, 6-months follow up.
  Used to provide an overall rating of the OCD severity. Clinician-rated. Range: 1-7, lower scores mean better outcome.
Clinical Global Impression - Improvement (CGI-I) | Post treatment (week 12), 3-months follow-up, 6-months follow up.
  Used to assess global improvement. Clinician-rated. Range: 1-7, lower scores mean better outcome.
Treatment response and remission | Post treatment (week 12), 3-months follow-up, 6-months follow up.
  Treatment response will be defined as at least 35% reduction on the CY-BOCS and a CGI-I score of 1 (very much improved) or 2 (much improved). Remission will be defined as a score of less than or equal to 12 on the CY-BOCS and a CGI-S rating of 1 (normal, not at all ill) or 2 (borderline mentally ill).
Children's Global Assessment Scale (CGAS) | Baseline (week 0), post treatment (week 12), 3-months follow-up, 6-months follow up.
  The CGAS is a single item 1-100 scale that integrates psychological, social, and academic functioning in children as a measure of psychiatric disturbance. Higher scores mean better outcome. It will be used in this trial to provide an assessor-rated opinion of global improvement (not restricted to OCD symptoms).
Obsessive-Compulsive Inventory - Child version - revised (OCI-CV-R) | Baseline (week 0), during treatment (week 3, week 6, week 9), post treatment (week 12), 3-months follow-up, 6-months follow up.
  The OCI-CV-R is an 18-item self-reported measure of OCD symptoms. Each item is scored on a 3-point scale (0=never, 1=sometimes, 2=always). The OCI-CV-R generates a total score ranging from 0-36 points and five sub-scores (doubting/checking, obsessing, washing, ordering, and neutralizing), with higher scores indicating greater OCD symptom severity.
Children's Obsessive-Compulsive Inventory-Revised-Parent version (ChOCI-R-P) | Baseline (week 0), during treatment (week 3, week 6, week 9), post treatment (week 12), 3-months follow-up, 6-months follow up.
  The ChOCI-R-P is a parent-rated measure of OCD symptom severity that includes a checklist and a severity rating with 12 items, yielding a total score of 0-48 with higher scores indicating greater OCD symptom severity.
Generalized Anxiety Disorder - 7 item scale (GAD-7) | Baseline (week 0), post treatment (week 12), 3-months follow-up, 6-months follow up.
  The GAD-7 is a measure of anxiety rated by the child/adolescent. It consists of 7 items and each item is rated from 0=not at all to 3=almost every day, yielding a total score of 0-21. Lower scores mean better outcome.
Child Health Utility 9D (CHU9D) | Baseline (week 0), post treatment (week 12), 3-months follow-up, 6-months follow up.
  The CHU9D is a 9-item measure of quality of life rated by the child/adolescent. Each item is scored from 1 to 5, assessing children's functioning "today" across domains of worry, sadness, pain, tiredness, annoyance, school, sleep, daily routine and activities. Scores are converted to utility weights using a scoring algorithm. Weights range between 0 (denoting the health state "dead") and 1 (denoting the health state "perfect health"). Weights are then used to estimate quality adjusted life years (QALY) to be used in the health economic evaluation.
Trimbos/iMTA Questionnaire for Costs associated with Psychiatric Illness (TiC-P) | Baseline (week 0), post treatment (week 12), 3-months follow-up, 6-months follow up.
  The TiC-P will be used to assess healthcare and societal resource use for the health economic evaluation. The questionnaire includes items on healthcare resource use (e.g., healthcare visits), supportive resources (e.g., private tutoring), medications, prescription-free drugs, school absenteeism, academic productivity loss, and parental productivity loss and is frequently used in health economic studies. The TiC-P version used in the study has been adapted by the research team for the use among young people and parents and used in previous trials. No scores as such are available for this measure. Parent rated.
Patient Exposure/Relaxation Adherence Scale (PEAS/PRAS) | During treatment (week 3, week 6, week 9), post treatment (week 12), 3-months follow-up.
  The PEAS/PRAS is a self-rated 3-item measure of patient adherence to exposure with response prevention (PEAS) with 3 items rated from 0 to 6, yielding a total score of 0-18, where higher scores indicate greater adherence. For the current trial, the measure will be administered as a self- rated version in the I-ERP group. A corresponding version (PRAS) has been developed by the research team and will be administered to participants in the control group to assess adherence to I-SM intervention.
  The PEAS/PRAS is a 3-item measure of patient adherence to exposure and response prevention (PEAS) or relaxation training (PRAS). The PEAS/PRAS is one single measure but it is adapted to each of the two arms. The PEAS/PRAS has 3 items rated from 0 to 6, yielding a total score of 0-18. Higher scores mean better outcome. For the current trial, the PEAS will be administered as a self-rated version in the I-ERP group and the PRAS will be administered as a self-rated version in the I-SM group.
Treatment preference | Baseline (week 0), post treatment (week 12).
  Two items will be administered to both the participant and the parent to assess treatment format preference (i.e., if the participant/parent would have preferred to receive internet-delivered treatment or in-person treatment for his/her symptoms or if it does not matter), as well as how important the participant and parent believe it is to be able to choose which treatment format they receive (rated on a 5-point scale). The questionnaire has been developed by the research team.
Treatment Credibility and Expectancy Scale (TCES) | During treatment (week 3).
  The TCES will be administered to both the participant and the parent to assess the treatment credibility and expectancy of treatment outcome. The TCES includes 5 items rated from 0 to 10, yielding a total score of 0-40, where higher scores indicate higher credibility.
Working alliance inventory (WAI) | During treatment (week 3).
  The WAI is a measure of perceived working alliance with the therapist that includes 6 items rated from 1=never to 7=always, yielding a total score of 7-49. It will be administered to both the participant and the parent. Higher scores mean better working alliance.
Client Satisfaction Questionnaire (CSQ-8) | Post treatment (week 12), 3-months follow-up.
  The CSQ-8 is an 8-item measure of treatment satisfaction. Each item is rated from 1 to 4, yielding a total score of 9-36. Higher scores mean more satisfaction. It will be administered to both the participant and the parent.
Family Accommodation Scale - self-rated (FAS-SR) | Baseline (week 0), post treatment (week 12), 3-months follow-up, 6-months follow up.
  The FAS-SR is a measure of family accommodation that includes 19 items about family accommodation. For the purpose of this trial, the checklist with obsessions and compulsions has been excluded, since it is not included in the total severity score and overlaps with the checklist in the ChOCI-R-P. Each item is rated from 0=none/never to 4=every day, yielding a total score of 0-76. Higher scores are associated with greater levels of family accommodation.
Work and Social Adjustment Scale - youth (WSAS-Y) | Baseline (week 0), post treatment (week 12), 3-months follow-up, 6-months follow up.
  The WSAS-Y is a 5-item measure of functional impairment rated by the child/adolescent. Each item is rated from 0=not at all to 8=severely impaired, yielding a total score of 0-40. Lower scores mean better outcome.
Work and Social Adjustment Scale - parent version (WSAS-P) | Baseline (week 0), post treatment (week 12), 3-months follow-up, 6-months follow up.
  The WSAS-P is a 5-item measure of functional impairment rated by the parent. Each item is rated from 0=not at all to 8=severely impaired, yielding a total score of 0-40. Lower scores mean better outcome.
Short Mood and Feeling Questionnaire - child (SMFQ-C) + additional suicide item | Baseline (week 0), during treatment (week 3, week 6, week 9), post treatment (week 12), 3-months follow-up, 6-months follow up.
  The SMFQ-C is a measure of depressive symptoms rated by the child/adolescent. It consists of 13 items and each item is scored on a 3-point scale (0=not true, 1=sometimes, 2=true). The total score is derived by adding up the values for each 13 items, yielding a total score of 0-26 points. Lower scores mean better outcome. For this trial, an item has been added aimed to assess suicide risk.
Short Mood and Feeling Questionnaire - parent version (SMFQ-P) | Baseline (week 0), during treatment (week 3, week 6, week 9), post treatment (week 12), 3-months follow-up, 6-months follow up.
  The SMFQ-P is a measure of depressive symptoms rated by the parent. It consists of 13 items and each item is scored on a 3-point scale (0=not true, 1=sometimes, 2=true). The total score is derived by adding up the values for each 13 items, yielding a total score of 0-26 points. Lower scores mean better outcome.

OTHER OUTCOMES:
Demographic data - clinician-entered | Baseline (week 0).
  Following the inclusion assessment, the assessor enters baseline information into the trial database. This includes information on e.g., age, primary responsible caregiver assisting during the treatment, general cognitive ability, comorbid diagnoses, distance to the clinic in kilometres, age of OCD onset, history of suicide attempt, family history of OCD and ASD, family history of other psychiatric disorders, current medication for ASD, OCD or other psychiatric disorder, and previous psychological treatment for OCD or other psychiatric disorders.
Demographic data - parent-reported | Baseline (week 0).
  At baseline, the parent/caregiver will answer a questionnaire designed by the research team asking about e.g., the caregiver's relation to the child, who the child lives with, the child's sex and gender, number of siblings, the caregivers' educational level, the caregivers' occupation, the country in which the child and caregivers were born, how the caregiver learned about the trial, and if the child has been in previous contact with health care services due to her/his OCD or other psychiatric symptoms.
Comorbid psychiatric disorders | Baseline (week 0).
  Psychiatric diagnoses at baseline will be based on DSM diagnostic criteria. OCD, and other obsessive-compulsive-related comorbidities will be evaluated via a semi-structured interview based on the Structured Clinical Interview for DSM-IV (SCID-IV), adapted to align with the more recent DSM-5 criteria. The presence of other psychiatric comorbidities will be assessed with the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).
Social Communication Questionnaire (SCQ) | Baseline (week 0).
  The SCQ is a parent-rated measure of autistic symptoms that includes 40 items, yielding a total score of 0-40.
IQ estimate | Baseline (week 0).
  Two subtests, matrix reasoning and similarities, from the WISC-V or WAIS-IV will be used to provide an estimate of full IQ.
Concurrent interventions | Post treatment (week 12), 3-months follow-up, 6-months follow up.
  To assess what other treatments the child/adolescent is accessing during the trial period, the family is interviewed by the assessor at post-treatment and subsequent follow-ups. This includes questions about medications (type, dose, indication, and time period) and psychological treatment (type, number of sessions, indication, and time period).
Adverse events | During treatment (week 6), post treatment (week 12), 3-months follow-up, 6-months follow-up.
  A questionnaire will be administered to systematically assess adverse events at mid-treatment, post-treatment, 3-month follow-up, and 6-month follow-up. The questionnaire is developed by the research team and includes a checklist with expected adverse events based on previous trials as well as a free text box where other, not listed adverse events can be registered.
School absenteeism - clinician | Baseline (week 0), post treatment (week 12), 3-months follow-up, 6-months follow up.
  The assessor will evaluate school absenteeism during the past month at all assessment points. The assessor will ask the participant and the caregiver if the participant has full, partial or no school attendance (i.e., school drop-out).
BASS platform usage data | Post treatment (week 12), 3-months follow-up.
  Usage data will be extracted from the BASS platform and entered into the trial database. These data are collected manually for each participant, including number of logins, number of messages sent to the therapist, and the name of the therapist.
Therapist time | Post treatment (week 12).
  The therapist time spent on each participant will be logged.
Completed modules | Post treatment (week 12).
  Descriptive statistics on the proportion of individuals in each group having completed at least 4 modules will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: David Mataix-Cols, Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Forskningsmottagning barn- och ungdomspsykiatri Lund, Lund, Skåne County
  - Child and Adolescent Psychiatry Research Center, Stockholm, Stockholm County
  - BUP Specialmottagning, Gothenburg, Västra Götalandsregionen

IPD SHARING:
Plan to Share IPD: No